CLINICAL TRIAL: NCT05174806
Title: A Randomized, Open Label, Controlled, Phase 2, Multi-Center Study to Assess Safety, Tolerability and Efficacy of Adjunctive Treatment With Topically Applied MBN-101 (Pravibismane Topical Suspension) in Subjects With Moderate Diabetic Foot Infection (DFI)
Brief Title: Multi-center Study to Assess Safety, Tolerability and Efficacy of Topical Pravibismane in Moderate DFI Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Microbion Corporation (Industry)
Collaborators: CUBRC (Unknown); National Medical Research Council (NMRC), Singapore (Other Government); MTEC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBN-101-203
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Infection; Diabetic Foot
Keywords: Amputation; DFI; Wound closure; Diabetic Foot Infection; Pravibismane; Clinical Cure; Safety and tolerability
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Topical Pravibismane (MBN-101) versus Standard of Care (SOC); 2:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical Pravibismane (MBN-101) (Experimental): Topical pravibismane (MBN-101) at a dose of 2.5 mg/mL will be applied directly to the infected wound and covered with an appropriate non-antimicrobial dressing. Dosing will occur 3 times per week for the 12 weeks of treatment.
  Interventions: Drug: Topical Pravibismane
- Standard of Care (Other): Standard of care treatment without administration of any topical drugs.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Topical Pravibismane — Topical Pravibismane
  Other Names: MBN-101
  Arms: Topical Pravibismane (MBN-101)
Other: Standard of Care — Standard of care treatment without investigational topical pravibismane (MBN-101) or other topical antibiotics.
  Other Names: SOC comparator
  Arms: Standard of Care

SUMMARY:
This is a randomized, open label, controlled, multi-center study to assess safety, tolerability, and efficacy of adjunctive treatment with topically applied pravibismane (MBN-101) in patients with moderate diabetic foot infections. Patients will be randomized in a 2:1 ratio (MBN-101:standard of care). Topical pravibismane (MBN-101) will be applied three times per week for up to 12 weeks. All patients will receive systemic antibiotic treatment for a least a portion of that period. Randomization will be stratified by site.

DETAILED DESCRIPTION:
This is a randomized, open label, controlled, multi-center study. Patients with diabetes mellitus (either type 1 or 2) and an infected wound of the foot with an International Working Group Diabetic Foot (IWGDF) severity rating of moderate will be eligible for the trial after meeting all inclusion criteria and none of the exclusion criteria.

Patients (n = 54) will be randomized in a 2:1 ratio (MBN-101: standard of care). Randomization will be stratified by site.

Patients randomized to the MBN-101 arm will be treated in an outpatient facility 3 times per week for the first 2 weeks. During each of the subsequent 10 weeks, patients will be treated once per week at the outpatient clinic and will be provided with enough MBN-101 for 2 additional days of treatment for self administration at home with or without the assistance of a caregiver. The duration between each dose should be greater than 24 hours, yet not exceed 72 hours for each of the 12 treatment weeks. Patients randomized to the standard of care arm will follow the same schedule (i.e., inclusive of wound dressing changes), though will not be treated with MBN-101.

All subjects will initially receive systemic antibiotic treatment and undergo appropriate sharp debridement at baseline and then as directed by the treating physician through the 12-week treatment period, yet part of the standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has diabetes mellitus, according to the American Diabetes Association (ADA) criteria.
* Has a skin ulcer located on or distal to the malleolus that is ≥ 4 weeks that is clinically documented, and presents with clinical manifestations of a moderate infection (i.e. erythema extending ≥ 2.0 cm from the wound margin), and not requiring hospitalization.
* Has received no more than 36 hours of antibiotic therapy for the moderately infected ulcer prior to enrollment or there is clinical and/or microbiological evidence of failure of antibiotic treatment for the treatment of the moderately infected ulcer.
* Has documented adequate arterial perfusion in the affected limb by biphasic or triphasic Doppler wave forms, a toe brachial index (TBI) ≥0.75, or an ankle brachial index (ABI) of >0.9).
* Has read and signed the Informed Consent Form (ICF) after the nature of the study has been fully explained.

Exclusion Criteria:

* Has proven or highly suspected, involvement of bone (i.e., osteomyelitis).
* Has an ulcer due to Charcot arthropathy.
* Has more than one concurrent, infected, diabetic foot wound on the study limb.
* Is unwilling or unable to attend clinic visits and keep research appointments.
* Is unwilling or unable to adhere to the systemic antibiotic treatment prescribed.
* Is unwilling or unable to adhere to proper pressure off-loading of the foot wound (when needed) from enrollment through EOS as directed by the treating physician.
* Has an untreated, uncontrolled, or poorly managed immunosuppressive and or autoimmune disorder.
* Plans to use any topical antibiotics, herbals remedies (e.g., honey), alternative medicines or antimicrobials, either directly or by dressings on their infected DFU at any time from enrollment through the EOS visit.
* Plans to receive treatment with larvae (maggots) for their infected DFU at any time from enrollment through the EOS visit.
* Plans to receive treatment with advanced cellular therapies (e.g., Platelet-derived growth factor (PDGF), Cellular Tissue Products (CTP), granulocyte colony-stimulating factor (G CSF)) for their infected DFU at any time from enrollment through the EOS visit.
* History of major medical noncompliance.
* Any condition that has required treatment with any other bismuth containing compound within 2 weeks prior to enrollment through EOS visit (i.e., Kaopectate or Pepto-Bismol, including topical applications such as Xeroform).
* Plans to receive treatment with Hyperbaric oxygen therapy (HBOT) or topical negative pressure wound therapy (NPWT) for their infected DFU at any time from enrollment through the EOS visit.
* Glycated hemoglobin >12%.
* Has a serum creatinine, ALT, AST or Alkaline Phosphatase >3 times the upper limit of the normal range of the local testing laboratory.
* End stage renal disease requiring dialysis.
* Has an absolute neutrophil count <1000.
* Has participated in an investigational trial to evaluate pharmaceuticals or biologics either concurrently or within the past 30 days.
* Will undergo a planned surgical therapy beyond standard bedside debridement or incision and drainage, to treat the DFI after enrollment.
* Has a known allergy to bismuth and/or MBN-101 excipients (methylcellulose, Tween 80 (polysorbate 80)).
* Is immunocompromised and not well-managed due to illness [human immunodeficiency virus (HIV), autoimmune disease] or organ transplant.
* Has a history of any type of cancer (excluding non-melanoma localized skin cancer or completely excised and cured carcinoma-in-situ of uterine cervix) unless the subject has been free of cancer for > 5 years.
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures.
* Active alcohol abuse (> 14 drinks per week over the last 3 months) or substance abuse (current use of cocaine, heroin, or methamphetamines) or if drug or alcohol use will interfere with visits in clinic in the opinion of the investigator.
* Has other medical condition(s) which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events | 12 weeks
  Safety and tolerability

SECONDARY OUTCOMES:
Proportion of subjects with complete wound closure | 12 weeks
  Effect of MBN-101 suspension on wound healing
Proportion of subjects with a clinical cure of infection | 12 weeks
  Effect of MBN-101 suspension on resolution of infection
Proportion of subjects undergoing lower-extremity amputation | 12 weeks
  Effect of topical pravibismane (MBN-101) suspension on the incidence of lower level extremity amputations

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Limb Preservation Platform, Inc., Fresno, California
  - Parkland Comprehensive Wound Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center University Wound Care Clinic, Dallas, Texas
  - University of Texas Southwestern Medical Center William P. Clements Jr. University Hospital, Dallas, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Bio-X-Cell Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No